CLINICAL TRIAL: NCT05216796
Title: Diet Intervention to Promote Liver and Brain Health in Adults With Non-alcoholic Fatty Liver Disease
Brief Title: Healthy Liver - Healthy Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Andreana P. Haley, Professor in Clinical Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002189
Record Dates: First submitted 2021-12-30; First posted 2022-02-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome; Non-Alcoholic Fatty Liver Disease; NAFLD; Pre-diabetes
Keywords: Neuroimaging; Liver; Low-carbohydrate; Diet
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: The investigators will employ a block randomization (n=10) between groups feeding trial where 100 participants will be assigned to receive either low-carbohydrate (LoCHO) or low-calorie (LoCAL) control diet for up to 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate diet (Experimental): Participants assigned to the Low-carbohydrate diet will be instructed to limit carbohydrate intake to <30 g/d.
  Interventions: Behavioral: Diet Intervention
- Low-calorie diet (Active Comparator): Participants assigned to the Low-calorie diet will be instructed to reduce their energy intake to match the LoCHO block (we are predicting ~1200 kcal/d for women and ~1500 kcal/d for men, following current recommendations for treatment of NAFLD).
  Interventions: Behavioral: Diet Intervention

INTERVENTIONS:
Behavioral: Diet Intervention — Meal will be prepared and delivered by SNAP Kitchen, which has 7 locations in Austin and offers 20+ options for low-carbohydrate and low-calorie meals, each meal available in different sizes varying in energy intake. Meals will be entered into the Nutrition Data System for Research (NDS-R) software to confirm low-calorie profile. Meals will be delivered to participants' homes twice a week.

SUMMARY:
People with liver disease report difficulties with attention and problem-solving skills. Diet plays an important role in the development of liver disease and/or pre-diabetes. The purpose of this study is to examine whether participation in a brief diet intervention (up to 3 weeks) can improve brain and liver health and function.

DETAILED DESCRIPTION:
The importance of liver function for brain and cognitive health is undeniable. Specifically, adults with chronic liver diseases such as non-alcoholic fatty liver disease (NAFLD), a factor of metabolic syndrome (MetS), experience a range of symptoms including problems with attention, problem solving skills and executive function. Importantly, diet plays a role in the development of NAFLD. The investigators propose to be the first to demonstrate that Metabolic syndrome-related brain vulnerability, in the form of elevated free cerebral glutamate, is related to hepatic triglyceride level, through experimental manipulation of liver fat and multiorgan imaging. The investigators seek to improve liver health by altering diet content in a block randomized feeding trial. The investigators selected a low-carbohydrate (<30 g/d) diet (LoCHO) to reduce liver fat and a low-calorie (LoCAL) diet as a control for weight loss. The investigators hypothesize that LoCHO diet will improve cognitive performance by improving liver health and thus, brain health. This work may provide a way to support brain function in MetS and delay cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age
* English speakers
* show a minimum of 5% hepatic triglyceride level on liver imaging
* have not taken part in a weight loss/dietary intervention within 6 months
* not currently adhering to a low-carbohydrate diet (e.g., Atkins, Paleo)

Exclusion Criteria:

* younger than 40 years of age
* have a history of neurological disease (e.g. stroke, seizure disorder)
* psychiatric illness (e.g. schizophrenia, bipolar disorder)
* harmful alcohol use (AUDIT-C score >5)
* morbid obesity (BMI>40)
* MRI contraindications

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Decrease in Liver Fat | Liver fat will be measured at baseline (week 0) and after at least 2 weeks (up to 3 weeks) on the designated diet. The liver 1H MRS scans will happen during Visit 3 (baseline) and Visit 4 (at least 2 weeks on the diet).
  Hepatic triglyceride level will be assessed using liver 1H MRS.
Decrease in cerebral gluatamate | Cerebral glutamate will be measured at baseline (week 0) and after at least 2 weeks (up to 3 weeks) on the designated diet. The brain 1H MRS scans will happen during Visit 3 (baseline) and Visit 4 (at least 2 weeks on the diet).
  Cerebral glutamate levels will be measured using 1H MRS.

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Haley, PhD, Principal Investigator — Department of Psychology, University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Browning JD, Baker JA, Rogers T, Davis J, Satapati S, Burgess SC. Short-term weight loss and hepatic triglyceride reduction: evidence of a metabolic advantage with dietary carbohydrate restriction. Am J Clin Nutr. 2011 May;93(5):1048-52. doi: 10.3945/ajcn.110.007674. Epub 2011 Mar 2. PMID 21367948
- [Background] Ervin RB. Prevalence of metabolic syndrome among adults 20 years of age and over, by sex, age, race and ethnicity, and body mass index: United States, 2003-2006. Natl Health Stat Report. 2009 May 5;(13):1-7. PMID 19634296
- [Background] Haley AP, Gonzales MM, Tarumi T, Tanaka H. Subclinical vascular disease and cerebral glutamate elevation in metabolic syndrome. Metab Brain Dis. 2012 Dec;27(4):513-20. doi: 10.1007/s11011-012-9306-x. Epub 2012 May 3. PMID 22552897
- [Background] Oh R, Gilani B, Uppaluri KR. Low-Carbohydrate Diet. 2023 Aug 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537084/ PMID 30725769
- [Background] Crabb DW, Im GY, Szabo G, Mellinger JL, Lucey MR. Diagnosis and Treatment of Alcohol-Associated Liver Diseases: 2019 Practice Guidance From the American Association for the Study of Liver Diseases. Hepatology. 2020 Jan;71(1):306-333. doi: 10.1002/hep.30866. No abstract available. PMID 31314133